CLINICAL TRIAL: NCT00875121
Title: Peer Interactions and Food Are Substitutable in Youth
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Sarah-Jeanne Salvy, Ph.D., University at Buffalo
Other Study IDs: DB#2220; 1R01HD057190-01A1 (NIH)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-04

CONDITIONS: Activity Choices; Caloric Intake; Social Time
Keywords: Food reinforcement; social reinforcers; overweight; children
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
This study examines the effects of increasing the cost of social interactions and food on overweight and non-overweight youth. Using a computerized operant task youth will earn points exchangeable for food and social activity.

The investigators predict that both overweight and non-overweight children will substitute food for interactions with an unfamiliar peer when this alternative is made expensive. Also, the investigators predict that both overweight and lean participants will defend their choice to spend time with a friend even when this alternative is made expensive.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 9-11
* Children must have a BMI equal to or greater than 15th percentile for their age
* Children must report at least a moderate liking of the study foods

Exclusion Criteria:

* Children should not have any food allergies
* Children should not have any dietary restraint
* Children should not a cold or upper respiratory distress
* Children should not have any psychopathology
* Children should not have any developmental disabilities
* Children should not be taking any medications that could influence their sense of smell and taste and activity level

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Boys and girls ages 9-11.
Sampling Method: Probability Sample
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Caloric Intake
Social Time

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Salvy, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Division of Behavioral Medicine, Buffalo, New York, United States